CLINICAL TRIAL: NCT06201052
Title: The Influence of Physical Exercise on Chosen Parameters of the Immune System, Prooxidant-Antioxidant Balance, and Iron Metabolism in Football Players With Various Training Levels
Brief Title: Impact of Exercise on Immune System and Metabolism in Football Players
Acronym: IEISM
Status: Completed | Type: Observational
Sponsor: Poznan University of Physical Education (Other)
Collaborators: Nicolaus Copernicus University (Other)
Responsible Party: Principal Investigator, Joanna Ostapiuk-Karolczuk, Principal Investigator, Poznan University of Physical Education
Other Study IDs: 382/2017
Record Dates: First submitted 2023-12-30; First posted 2024-01-11 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Healthy
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Junior: Junior soccer players 19 male, average training experience: 8 years
  Interventions: Other: Exercise test
- Senior: Senior Soccer players 21 male, average training experience: 16 years
  Interventions: Other: Exercise test

INTERVENTIONS:
Other: Exercise test — Beep Test for measuring aerobic power

SUMMARY:
Physical exercise, especially of high intensity, is a significant burden to the athlete's body. It should be emphasized that achieving high results in competitive sports requires significant, sometimes extreme, exercise loads during training, which may result in homeostasis disorders, adversely affecting athletes' fitness. Intense and prolonged physical exercise elevates reactive oxygen species, potentially impacting immune function. The mechanism, particularly in high-intensity activities, remains incompletely understood. Excessive oxygen radicals may induce metabolic changes, causing rapid erythrocyte damage and elevated redox-active free iron. This iron increase can be harmful, increasing oxidative stress and immune system activation. The sustained negative impact that may be observed even during post-workout recovery needs further exploration.

"This study aims to explain the impact of an intense exercise test on the immune system, pro-antioxidant balance, and iron metabolism in athletes with varying training levels. The primary questions it seeks to address are:

1. How do athletes' experience and training background influence the immune system's response, pro-antioxidant balance, and iron regulation?
2. Can the level of adaptation to physical exercise (training status) affect the rate of regeneration and the time required to return to pre-exercise homeostasis?"

DETAILED DESCRIPTION:
The study included 40 football players (19 juniors and 21 seniors). The average training experience for junior players was 8.37 years, and for the senior group, it was 16.4 years. All athletes underwent the Multistage 20-meter shuttle run test (Beep Test). Players were informed about the test procedures and additionally motivated by the trainer to exert maximum effort. Each attempt was preceded by a warm-up, consisting of a 5-minute low-intensity jog. The Beep Test was supervised by the Team trainer using a program as a monitoring tool to examine changes in the level of cardio-respiratory fitness across all age groups. Blood samples were collected at rest, before the exercise test, then 1 minute after the end of the exercise test, after 3 hours of recovery, and finally, after 24 hours. Blood was drawn from the antecubital vein, with 12 ml collected each time.

ELIGIBILITY:
Inclusion Criteria:

* Competitive football training for at least 3 years
* Male
* Not taking any medications throughout the study
* Provide voluntary consent for participation in the study

Exclusion Criteria:

* Any healthy problems

Ages: 22 Years to 37 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Forty healthy football players, aged from 22 to 37 years. The average training experience for junior players was 8 years and 16 for the senior group.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Changes in iron level | At rest (before the exercise test), 1 minute after the end of the test, after 3 hours, and 24 hours of recovery.
  marker of iron management
Changes in UIBC (unsaturated iron-binding capacity) | At rest (before the exercise test), 1 minute after the end of the test, after 3 hours, and 24 hours of recovery.
  marker of iron management
Changes in TIBC (total iron-binding capacity) | At rest (before the exercise test), 1 minute after the end of the test, after 3 hours, and 24 hours of recovery.
  marker of iron management
Changes in hepcidin | At rest (before the exercise test), 1 minute after the end of the test, after 3 hours, and 24 hours of recovery.
  marker of iron management
Changes in lactoferrin | At rest (before the exercise test), 1 minute after the end of the test, after 3 hours, and 24 hours of recovery.
  marker of iron management
Changes in IL-6 (interleukin-6) | At rest (before the exercise test), 1 minute after the end of the test, after 3 hours, and 24 hours of recovery.
  marker of immune system
Changes in IL-10 (interleukin-10) | At rest (before the exercise test), 1 minute after the end of the test, after 3 hours, and 24 hours of recovery.
  marker of immune system
Changes in TNF-α (tumor necrosis factor-alpha) | At rest (before the exercise test), 1 minute after the end of the test, after 3 hours, and 24 hours of recovery.
  marker of immune response
Changes in tryptophan | At rest (before the exercise test), 1 minute after the end of the test, after 3 hours, and 24 hours of recovery.
  marker of immune response
Changes in IGF-1 (insulin-like growth factor 1) | At rest (before the exercise test), 1 minute after the end of the test, after 3 hours, and 24 hours of recovery.
  marker of hormonal response
Changes in testosterone | At rest (before the exercise test), 1 minute after the end of the test, after 3 hours, and 24 hours of recovery.
  marker of hormonal response
Changes in cortisol | At rest (before the exercise test), 1 minute after the end of the test, after 3 hours, and 24 hours of recovery.
  marker of hormonal response
Changes in serotonin | At rest (before the exercise test), 1 minute after the end of the test, after 3 hours, and 24 hours of recovery.
  marker of neurohormonal response
Changes in myoglobin | At rest (before the exercise test), 1 minute after the end of the test, after 3 hours, and 24 hours of recovery.
  marker of muscle damage

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Ostapiuk-Karolczuk, Ph.D., Principal Investigator — Poznan University of Physical Education
Locations (1):
- Poznań University of Physical Education, Poznan, Poland

IPD SHARING:
Plan to Share IPD: No